CLINICAL TRIAL: NCT02414438
Title: Establishing the Clinical Utility of First StepDx PLUS and NextStepDx PLUS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Lineagen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01-LIN-2014
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Intellectual Disability; Developmental Delay
MeSH Terms: conditions — Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Current Practice Arm (No Intervention): Physicians follow current care procedures
- FirstStep and NextStep Information (Experimental): Providers receive informational webinar regarding FirstStepDx PLUS and NextStepDx PLUS between rounds and are able to order test results in Round 2
  Interventions: Other: FirstStepDX PLUS and NextStepDX PLUS Webinar
- FirstStep and NextStep Results (Experimental): Providers receive informational webinar regarding FirstStepDx PLUS and NextStepDx PLUS between rounds and are specifically prompted to order test results in Round 2
  Interventions: Other: FirstStepDX PLUS and NextStepDX PLUS Webinar; Other: FirstStepDX PLUS and NextStepDX PLUS Test Results

INTERVENTIONS:
Other: FirstStepDX PLUS and NextStepDX PLUS Webinar — A pre-recorded 20-minute webinar on FirstStepDX PLUS and NextStepDX PLUS
  Arms: FirstStep and NextStep Information; FirstStep and NextStep Results
Other: FirstStepDX PLUS and NextStepDX PLUS Test Results — Physicians receive a prompt to order and download FirstStepDX PLUS and NextStepDX PLUS Test Results
  Arms: FirstStep and NextStep Results

SUMMARY:
The study uses a randomized controlled study design of pediatric neurologists and developmental pediatricians and front-line (primary care) pediatricians to determine if use of FirstStepDx PLUS and Next StepDx PLUS are associated with higher clinical quality, less variability in clinical practice, and lower costs from decreased resource utilization. The Clinical Performance and Value Vignettes (CPV) used in this study simulate a clinical encounter for individuals with an atypical phenotype and clinical presentation indicative of a possible genetic disorder. We will measure the difference in combined diagnostic and treatment CPV® domain score post-intervention versus baseline comparing intervention and control groups

DETAILED DESCRIPTION:
The study is an interventional longitudinal study design of physician practice. 225 specialist and general pediatricians without previous exposure to FirstStepDx PLUS or NextStepDx PLUS will be selected from a nationally representative list of approximately 25,000 board-certified pediatricians and 5,000 specialists. These physicians will be randomized into one of three arms: to receive information regarding FirstStepDx PLUS ("Intervention A"), to receive information about FirstStepDx PLUS and NextStepDx PLUS ("Intervention B") for use in clinical practice, and controls not receiving any intervention. Specifically we will test the hypotheses:

1. Clinical practice, specifically decisions around treatment of individuals with disorders postnatal development including DD, ASD, and ID will vary widely among all physician types. This documentation of variation in practice will demonstrate the need for a new diagnostic service that FirstStepDx PLUS and NextStepDx PLUS would fulfill
2. FirstStepDx PLUS and NextStepDx PLUS will improve the quality and appropriateness of care and therapeutic plans, as measured by the number of physicians that correctly act on the results of the assay

A Physician Questionnaire will be administered to all physicians. This questionnaire will assess physician, patient and practice characteristics. Data gathered from this set of questions will become part of the baseline (pre-intervention) assessment and used for analysis. At the baseline assessment, Clinical Performance and Value (CPVs) Vignettes, a validated tool to measure physician performance and behavior will be used. CPV vignettes have been used to establish clinical utility in the molecular diagnostic space.

The CPV vignettes used in this study will simulate a clinical encounter for a patient with an atypical clinical presentation indicative of a possible genetic developmental disorder. Each physician will provide open-ended responses regarding clinical care. These responses are scored in five domains (taking a medical history, performing a physical examination, ordering appropriate tests, making a diagnosis and prescribing treatment against explicit evidence and criteria as determined by the literature and by expert physicians. Results are presented as percentage correct controlling for primacy effects using case within pair randomization. Each case will take approximately 15-20 minutes to complete. All case responses will be completed electronically online and confidential. No physician or practice names are used when reporting the results of the study.

The CPVs will be randomly assigned to physicians for each to complete 3 CPVs™ (one from each type). Each of the CPVs will be scored by physicians for changes in clinical practice including treatment changes, frequency of follow up, laboratory tests and imaging studies ordered - see for scoring sheet.

The objective of this study is to assess how FirstStepDx PLUS (and NextStepDx PLUS) testing affects the variability of clinical practice and resultant impact.

Primary Endpoint Differences in CPV diagnosis/treatment domain score post-intervention versus baseline for the intervention and control group physicians).

Secondary Endpoints

* Difference in utilization of appropriate treatment including indicated versus unnecessary therapy pre- and post-intervention between intervention and control groups
* Difference in utilization of laboratory testing such as fluorescence in situ hybridization (FISH) analyses, global assessment, and utilization of other laboratory tests pre- and post-intervention, between intervention and control groups
* Difference in overall Clinical Performance and Value Vignettes (CPV®) scores post-intervention versus baseline between intervention and control groups

ELIGIBILITY:
Inclusion Criteria:

1. Provide consent to participate in the study
2. Currently practicing board-certified physician in the following specialty areas:

   1. Pediatric neurologists
   2. Developmental pediatricians
   3. General pediatricians
3. Have practiced as a board-certified physician for greater than 2 but less than 30 years.
4. English-speaking
5. Community / non-academic based practice setting
6. ≥30 pediatric patients under care annually
7. Access to the internet

Exclusion Criteria:

1. Not board certified in their respective area of care
2. Academic-based practice
3. Have previously used FirstStepDx PLUS and/or NextStepDx PLUS in their care delivery
4. Have practiced as a board-certified physician for less than 2 or greater than 30 years.
5. Follow <30 pediatric patients annually
6. Non-English speaking
7. Unable to access the internet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis and Treatment Score | 4 weeks
  Differences in CPV diagnosis/treatment domain score post-intervention versus baseline for the intervention and control group physicians).

SECONDARY OUTCOMES:
Overall CPV score | 4 weeks
  Differences in overall CPV score post-intervention versus baseline for the intervention and control group physicians).

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD PhD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, San Rafael, California, United States

REFERENCES:
- [Background] Peabody JW, Luck J, Glassman P, Jain S, Hansen J, Spell M, Lee M. Measuring the quality of physician practice by using clinical vignettes: a prospective validation study. Ann Intern Med. 2004 Nov 16;141(10):771-80. doi: 10.7326/0003-4819-141-10-200411160-00008. PMID 15545677